CLINICAL TRIAL: NCT04661475
Title: Dexmedetomidine Adjuvant Treatment for Depressed Patients Undergoing ECT: A Double Blind, Placebo Controlled, Randomized Feasibility Study Protocol
Brief Title: Dexmedetomidine Adjuvant Treatment for Depressed Patients Undergoing ECT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Mohammed Al Alawi, Principal Investigator, Dr Mohmmed Al Alawi Bsc, MD, MRCPsych, OMSBPsych, ARABPsych, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13/2020
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: .A double blind, placebo controlled, randomized Feasibility Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine adjunctive to ECT arm (Experimental)
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- Normal Saline adjunctive to ECT arm (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — ECT and anaesthetic treatment protocols will be determined by the local ECT services. ECT being given twice a week. The anesthetic induction agent of choice will usually be propofol, with thiopental permissible as an alternative. For safety reasons, any drug contraindicated to be given with DEX will be avoided. Especially the once known to decrease arterial pressure and heart rate excessively. Oral psychotropic medication to be continued by the patient's treating clinical team will remain unchanged where possible for at least the first 4 ECT treatments, and ideally until end of ECT. Eligible subjects will be allocated randomly to receive either 0.5µg/kg dexmedetomidine add on (diluted to 10 ml with 0.9% saline) at a steady rate of 1 ml/min, for 10 min.Participants in the two groups will receive DEX or Saline adjunct thrice weekly for 3 weeks.
  Arms: Dexmedetomidine adjunctive to ECT arm
Drug: Normal saline — while patients in the Control group will be infused with 10 ml of 0.9% saline at the same rate, over 10 minutes before anesthesia induction for ECT procedure.
  Arms: Normal Saline adjunctive to ECT arm

SUMMARY:
Major depressive disorder (MDD) is a highly prevalent and disabling condition for which the currently available treatments are not fully effective. Existing unmet needs include rapid onset of action and optimal management of concurrent agitation. Preliminary data support Dexmedetomidine as an antidepressant with fast onset of action, which would be especially helpful for patients experiencing treatment resistant depression, and agitation This trial will recruit 76 participants from the ECT waiting list at department of psychiatry and randomize them to either Dexmedetomidine infusion (0.5µg/kg/hr for 15 mins ) adjunct to ECT or Placebo adjunct to ECT( Saline) treatment arm added to standard anesthetic induction in depressed patients who have been prescribed ECT utilizing fixed randomization schedule that allocate subjects in to a 1:1 ratio between two arms.. Participants will receive ECT as described in the study schedule and as decided by their treating physician. Throughout the study, clinical, neuroimaging, molecular, and cognitive assessments will be conducted.

The trial aims to show that compared with Placebo adjunct to ECT( Saline) treatment, Dexmedetomidine infusion adjunctive treatment will lead to higher and faster response rate in depression, lesser number of ECT sessions required to achieve antidepressant response, less incidence of confusion post ECT and comparable incidence of side effects . This could lead to faster, more effective treatment for patient with depression

DETAILED DESCRIPTION:
Dexmedetomidine adjuvant treatment for depressed patients undergoing ECT. A double blind, placebo controlled, randomized Feasibility Study Protocol.

Introduction Major depressive disorder (MDD) is one of the most common mental illnesses, with lifetime prevalence around 7.2% (Lim et al., 2018). MDD has a detrimental impact on the quality of life and the ability to function of those affected by it and is considered one of the leading causes of disability worldwide (Vos et al., 2015). Moreover, MDD is associated with a significant disease burden for the affected individuals, their families and society at large (GBD 2015 DALYs and HALE Collaborators et al., 2016). By 2030, MDD is predicted to have the highest impact (i.e. most debilitating) among all conditions worldwide (Mathers et al., 2006). Although full remission is seen as the ultimate target for individuals suffering from MDD, existing evidence suggests that approximately two-thirds of MDD patients fail to attain or maintain full remission with the currently available antidepressant treatments (Trivedi et al., 2006). Individuals who do not have a satisfactory response to at least two different antidepressants at their adequate dose/duration of treatment are considered to be treatment-resistant depression (TRD) patients (Fava et al., 2003). TRD or difficult to treat depression (DTD) represents a clinical challenge, with a significant burden that is hard to estimate, as this condition is multi-episodic, often pervasive, with chronic and severe symptoms (Fekadu et al., 2018; Zhou et al., 2015).

Depression is a heterogenous disorder, both phenotypically and neurobiologically, with psychomotor agitation being a significant clinical challenge when treating individuals with this disabling condition (Fried et al., 2015). Another pragmatic challenge is the optimization of treatments for patients who exhibit concurrent subthreshold symptomatology of hypomania or mania. Although there are several guidelines available for the treatment of unipolar depression, bipolar depression and bipolar mania, specific treatments for depression with psychomotor agitation, depression with anxious- distress and depression with mixed features are scarce. Hence, there is a need for new therapeutic agents that could target this subset of depressed individuals.

Dexmedetomidine (DEX). DEX, (S)-4-[1-(2,3 dimethylphenyl)ethyl]-3H-imidazole], is a selective and potent α2-adrenergic receptor (α2-AR) agonist which was approved for the sedation of patients admitted to intensive care units (ICUs) by the FDA in 1999 (McCutcheon et al., 2006).

Mechanistic evidence of DEX antidepressant activity DEX Pharmacological characteristics {INSERT FIGURE 1} DEX is the S-enantiomer of the veterinary sedative: medetomidine. DEX is a highly selective α2-adrenoceptor agonist with an α2:α1 selectivity ratio of 1620:1 (Scott-Warren et al., 2015). DEX exerts its agonistic action on (A) subtype of α2 adrenoceptor; an activation of A subtype of α2 seems to lead to a protective effect against depression (Rivero et al., 2016; Schramm et al., 2001). Additionally, this activation appears to have analgesic and anxiolytic properties (Weerink et al., 2017). A recent comprehensive review noted that DEX has organ-protective effects, including neuroprotection, cardio-protection and renoprotection, through modulating gene expression, channel activation, transmitter release, and apoptotic and necrotic cell death. DEX shows protective effects in a variety of animal models of ischemia/reperfusion injury, including in the intestine, myocardial, renal, lung, cerebral and liver (Biccard et al., 2008; Wijeysundera et al., 2003).

DEX has been found to have anti-inflammatory properties and play a role in preventing the brain from stress response due to ischemic/reperfusion injury (Dahmani et al., 2005; Gu et al., 2011). Studies have demonstrated that sedation with DEX significantly decreases cytokine production, including IL-1p, TNF-[alpha], and IL-6, in critically ill patients and that DEX decreases the levels of TNF-[alpha], IL-1 and IL-6 to an even greater extent than propofol (Venn et al., 2001).

Following intravenous administration, DEX exhibits the following pharmacokinetic properties: a rapid distribution phase with a distribution half-life of approximately 6 minutes; a terminal elimination half-life of approximately 2 hours; and steady-state volume of distribution of approximately 118 liters. Clearance is estimated to be approximately 39 liters per hour. The mean body weight associated with this clearance estimate was 72 kg. DEX exhibits linear kinetics in the dosage range of 0.2 to 0.7 mg/kg/hr when administered by IV infusion for up to 24 hours (Weerink et al., 2017).

Preclinical Data on DEX antidepressant potential Moon et al. (2018) conducted the first animal study exploring the antidepressant effects of DEX on the depressive behaviors of sleep-deprived mice (Moon et al., 2018). The mice in this study were studied in 5 groups, with 10 mice in each group, as follows: control, sleep deprivation, sleep deprivation and 0.5 μg/ kg of DEX, sleep deprivation and 1 μg/kg, and sleep deprivation and 2 μg/kg DEX. Depressive behaviors were determined using the forced swimming and tail suspension tests (Holmes et al., 2005). In order to assess the effect of DEX on the expression of tyrosine hydroxylase (TH), 5-hydroxytryptamine (5-HT; serotonin), tryptophan hydroxylase (TPH) and D1 dopamine receptor, Western Blots and immunohistochemistry tests were run on mouse brain tissue. The sleep deprivation took 7 days in total, from day one, after the induction, DEX was injected into the mice once daily for 6 days, with dosing specific to the group allocation. After 6 days of DEX injections, depressive behaviors were assessed among the five groups and then brain tissues were examined. The results showed that sleep deprivation induced depressive behaviors in the form of increased latency to immobility in the forced swimming test and tail suspension test. Additionally, sleep deprived mice had decreased expressions of TPH, 5-HT, and D1 dopamine receptor, and increased TH expression. After 6 injections, DEX-alleviated depressive behaviors were evident through decreased latency to immobility, increased expressions of TPH, 5-HT, and D1 dopamine receptor, and decreased HT expression. The effects were statistically significant and incremental in a dose-dependent manner.

In another animal study conducted by Gao et al., DEX improved learning and memory impairment caused by ECT in depressed mice. DEX cognitive neuroprotection was achieved by suppressing excessive up-regulation of NR2B, a subunit of the NMDA receptor (Gao et al., 2016). Noteworthy, ketamine (another agent with rapid antidepressant effects) likely exerts its antidepressant properties through its antagonism of the NR2B-subunit-containing NMDA receptors (Gass et al., 2018). Therefore, one could suggest that DEX may exert its antidepressant action, at least in part, through modulation of NMDA receptors. Table 2 summarizes four preclinical animal studies postulating DEX antidepressant potential.

Clinical data on DEX A number of studies have shown showed positive outcomes following the use of DEX for the management of agitation among ICU patients, including a reduction in the number of cases of delirium, and shorter stays in ICU, which is likely due to an increased ease in moving off of mechanical ventilation, as well as an improvement in overall survival (Bougarel et al., 2011; Constantin et al., 2016; Dahmani et al., 2005; Ebert et al., 2000; Gao et al., 2016; Gass et al., 2018; Holmes et al., 2005; Ji et al., 2017; Jun et al., 2017; MacMillan et al., 1996; Moon et al., 2018; Venn et al., 2001; Weerink et al., 2017; Yuen et al., 2008).

DEX has been utilized by different specialties like anesthesiology, surgery, neurosurgery, and dentistry, for its sedative and anti-inflammatory potentials (Chandanwale et al., 2017). DEX has various clinical advantages, including induction of moderate sedation, a wide therapeutic index, the absence of infusion rates adaptation outside hepatic insufficiency and pronounced analgesic action (Reade et al., 2009). DEX is commonly used in an off-label manner in pediatric intensive care units (Baarslag et al., 2017). Additionally, DEX has proven to be an effective drug for MRI sedation, as well as the ambulatory sedation of pediatric population (Mason et al., 2008; Siddappa et al., 2011).

More recently, Yu et al. (2019) published the first study examining the efficacy of post-delivery DEX infusion in preventing postpartum blues or postpartum depressive symptoms (measured by Edinburgh Postnatal Depression Scale -EPDS), postpartum self-harm ideation (at postpartum days 7 and 42), pain symptoms and sleep problems. This study was a double-blind randomized placebo-controlled clinical trial, conducted at tertiary care university hospital in China. The subjects (n = 600) were women who underwent elective cesarean section under spinal anesthesia and accepted patient-controlled intravenous analgesia (PCIA). Participants were at least 18 years of age and class II according American Society of Anesthesiologists. Exclusion criteria included history of bipolar or psychotic disorder; suicidal state; allergies to a2-AR agonists; drug and/or alcohol abuse within the past 6 months; and use of another a2-AR agonist or a2-AR antagonist during the observation. Individuals assigned to the DEX group received 0.5 µg/kg intravenous DEX after delivery, at an infusion speed of 0.375 ml/kg per hour and infusion time of 20 minutes. The control group received 0.125 ml/kg intravenous 0.9% normal saline immediately after delivery at an infusion speed of 0.375 ml/kg per hour and infusion time of 20 minutes. The PCIA protocol for the control group consisted of 150 µg sufentanil diluted to 150 ml and administered at a continuous dose of 0.04 µg/kg per hour and a bolus dose of 2.0 µg, with a lockout of 8 minutes. DEX arm PCIA protocol was 150 µg sufentanil plus 150 µg DEX diluted to 150 ml, with the continuous dose of sufentanil 0.04 µg/kg per hour and DEX 0.04 µg/kg per hour, and a bolus dose of 2 µg, with a lockout of 8 minutes. The PCIA pump was stopped 48 hours postoperatively. All participants were monitored for pulse oxygen saturation, electrocardiogram, and noninvasive blood pressure for 48 hours after surgery. Participants were followed at 6, 24, and 48 hours for side effects and the status of sedation analgesia and slumber.

Antenatal and postnatal depressive symptoms were assessed with the Edinburgh Postnatal Depression Scale (EPDS), with an EPDS of 10 or higher indicating threshold for antenatal depressive symptoms. Sleep quality was assessed with the Insomnia Severity Index (ISI). After delivery, depressive symptoms EPDS and ISI were noted by blinded investigators by telephone at 7 and 42 days after delivery. If participant could not be contacted on 7 and 42 days, the investigator would try to reach them again by phone within 2 days. If participant was not contactable, they were deemed lost to follow-up. Sedation was assessed using the Ramsay sedation scores, recorded at 6, 24, and 48 hours after surgery. Postoperative analgesia was assessed using the numerical rating scale (NRS), recorded at 6, 24, and 48 hours after surgery. The quality of sleep was assessed with the ISI before surgery and on postpartum days 2, 7, and 42. The results showed good compliance, with 276 of 300 (92%) participants in the control group and 281 of 300 (93.67%) in the DEX group completing all follow up visits. There were no significant differences regarding demographic or clinical characteristics between the two groups, including significant antenatal depressive scores among DEX and control individuals (27.8% vs 30.1%, P = 0.55).

The incidence of PDS (EDPS score of ≥ 10) in the control group and DEX group were 16.3% and 5.7%, respectively, significantly lower among the individuals who were administered DEX (P <0.001). The EPDS score (mean and SD) at postpartum day 7 (1.93 ± 3.36 vs 4.23± 4.37, p<0.001) and at postpartum day 42 (1.99± 3.18 vs 4.68 ± 4.78, p<0.001) in the DEX group were also significantly lower than that observed in the control group. Logistic regression analysis showed that stress during pregnancy, antenatal depressive symptoms, life stress events, and domestic violence were risk factors for PDS. Notably, logistic analysis showed that the prophylactic use of DEX was a protective factor against PDS adjusted odds ratios (0.230; 95% CI: 0.104-0.510). Postpartum analgesia scores at 24 and 48 hours postpartum within the DEX group were significantly lower than that in the control group (P <0.001). The sleep score (ISI) at postpartum 48 hours in the DEX group was significantly better than that in the control group (P <0.001). Compared with the control group, the incidence of self-harm ideation in the DEX group significantly decreased at postpartum day 7 (4.0% vs 1.1%, P = 0.03) and day 42 (2.9% vs 0.4%, P = 0.04). No significant difference was observed in the incidence of nausea, vomiting, or dizziness between the control and the DEX group (1.07% vs 1.45%, P = 0.98; 2.85% vs 4.23%, P = 0.34; 10.68 vs 11.27, P = 0.83). Hypotension, bradycardia, hypoxemia, and respiratory depression were not observed in either of the two groups at 48 hours postpartum.

The impact of DEX on EPDS scores at day 42, showed an effect size of Cohen's D = 0.6 (Yu et al., 2019). This study seems to suggest promising results for the prophylactic effects of DEX against the emergence of postpartum depression. Ge Huang et al., 2020 reported a case of patient with resistant cancer pain and comorbid depressive illness who improved from mood and pain perspectives after treated with co-administration of DEX and morphine intrathecal. Depression was assessed by HAMD-6 before and after 1 week, one and three month of DEX addition to the regimen. The results showed positive changes in depressive symptoms and quality of life over the next 3 months.

No trials to date, however, have explored the efficacy of DEX for the treatment of individuals with a current episode of MDD.Taking together all existing pre-clinical and clinical data (despite their limitations) and the known pharmacological properties of DEX, we believe that there could be a potential use for DEX beyond its current use to manage agitation and to induce sedation in ICU settings, i.e., there seems to be a rationale for further exploration of the putative rapid antidepressant effects of DEX. The anti-agitation properties of DEX could be especially useful for individuals with depression accompanied by agitation or with mixed features. There is also potential for DEX to be used as a monotherapy when fast onset of action is required, as well as an alternative and/or as adjunctive therapy for other fast action interventions for MDD (ECT, rTMS).

Aims and Hypotheses The primary aim of the DEX-ECT study is to explore the effect of adjunctive DEX on response rate among a sample of depressed patients undergoing ECT using an RCT design with the hypothesis that adjunct DEX, compared with adjunct placebo (saline treatment), given prior to standard anesthesia will lead to a higher response rate. Secondary aims are to investigate the remission rate, tolerability and acceptability of adjunctive DEX. We hypothesize that DEX arm will show higher remission rate in depressive symptoms with no statistically significant difference in the rate of side effects during and post ECT between the two arms).

Design and study site A double blind, parallel group, placebo controlled, randomized feasibility trial will be conducted at, Department of Psychiatry, Queens University, Canada, over 6 week period. Enrolled patients will be randomized to DEX infusion (0.5µg/kg/hr for 15 mins ) adjunct to ECT or Placebo adjunct( Saline) treatment arm added to standard anesthetic induction in depressed patients who have been prescribed ECT utilizing fixed randomization schedule that allocate subjects in to a 1:1 ratio between two arms. Both subjects and outcome assessors will be blinded to the treatment arm to which participants are allocated. Given non- maleficence principle, the anesthetic team will be aware of treatment allocation, and should safety concern arise research investigators will be informed as well.

Allocation concealment, randomization All participants will be randomly allocated to the dexmedetomidine group (Dex group) or the control group (Normal Saline) using a computer-generated random number with a 1:1 allocation. An independent investigator, not involved in the clinical management or data collection, keep allocation data. The allocation details will be delivered in a sealed, opaque envelope in order to enable patients and assessors to remain blinded to group allocation. Prior to ECT, anesthesiologists who will not participate in data analysis will be informed about allocation, and the related data will be gathered during ECT by an independent staff blinded to treatment allocation. On the day of each treatment the anaesthetist. will open the package and prepare the injection away from the ECT team and patient to maintain their blinding. Patients will receive the same allocated study medication throughout their course of ECT. The allocation will not be revealed until final statistical analysis is completed. The final decision to end ECT will rest with the treating clinical team in consultation with the patient and the local ECT treatment team.

Sample Size Power estimates for continuous MADRS scores assumed a two-tailed alpha level of 0.05. Effect size estimate, Cohen's d=0.66 for DEX on post-partum depression symptoms scores was derived from previous study (Yu et al, 2019). A group of 76 patients randomly assigned in a 1:1 ratio (38 DEX versus 38 Placebo) will provide 80% power to detect a significant difference in the mean changes in MADRS scores between the two study arms. Since this is a feasibility study, 30 participants per each arm could be acceptable (Billingham, S. A., Whitehead, A. L., & Julious, S. A. (2013).

ELIGIBILITY:
Inclusion Criteria:

* -Male and female patients aging 18-70 years, with a DSM-5 diagnosis of MDD who will be commenced on ECT treatment by their treating psychiatrist.
* American Society of Anesthesiologists' (ASA) Physical Status class of I-II.
* Verbal IQ equivalent to 85 or greater and sufficiently fluent in English to validly complete neuropsychological testing.
* Provision of written informed consent before initiation of any study-related procedures.
* Eligible participants who have consented to standard ECT treatment for their mood disorder and are willing to accept randomization to either DEX+ECT or Placebo+ECT
* Subjects meeting criteria for Major Depressive Disorder (MDD) according to the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) currently in a Major Depressive Episode (MDE) as confirmed by the MINI International Neuropsychiatric Interview (MINI).
* A Montgomery-Åsberg Depression Rating Scale (MADRS) total score of ≥ 26 at screening and at randomization, with no more than 20% improvement between these two visits.
* Female subjects of childbearing potential must have a negative urine pregnancy test at enrolment (Visit 1) and be willing to use a reliable method of birth control (i.e., double-barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal ligation) during the study.
* Be able to understand and comply with the requirements of the study, as judged by the investigator(s).

Exclusion Criteria:

* -Prior or current substance abuse or dependence (except for caffeine or nicotine dependence) and/or recent history (last 12 months) of current alcohol abuse or dependence, as defined in DSM-5 criteria ("a problematic pattern of using alcohol or another substance that results in impairment in daily life or noticeable distress").
* A positive toxicology screen for drugs that are not prescribed and Alcohol Use Disorder
* Vascular Depression due to stroke, or MDD in the context of cancer diagnoses or other severe medical illnesses( SLE, MS etc)
* Unwilling to maintain current antidepressant regimen.
* Unwilling to discontinue any narcotic for a minimum of 5 drug half-lives prior to DEX infusion
* Pregnant, lactating, or of childbearing potential and not willing to use an approved method of contraception during the study.
* Evidence of clinically relevant disease, e.g., uncontrolled hypertension, hypotension, renal or hepatic impairment, significant coronary artery disease (myocardial infarct within a year prior to initial randomization), cerebrovascular disease, cardiac insufficiency, sick sinus syndrome, bradycardia, atrioventricular block of degree II and III, history of cerebrovascular accident, viral hepatitis B or C, acquired immunodeficiency syndrome.
* A clinical finding that is unstable or that, in the opinion of the investigator(s), would be negatively affected by the study medication or that would affect the study medication (e.g., diabetes mellitus, hypertension, unstable angina).
* Liver function tests AST and ALT three times the upper normal limit at screening.
* Uncorrected hypothyroidism or hyperthyroidism. Subjects needing a thyroid hormone supplement to treat hypothyroidism must have been on a stable dose of the medication for 30 days prior to enrolment (Visit 1).
* Clinically significant deviation from the reference range in clinical laboratory test results( of liver , renal , thyroid, complete blood count ) as judged by the investigator(s).
* ECG results considered clinically significant as determined by the investigator(s), or outside of normal range as per cardiologist analysis.
* History of seizure disorder, except febrile convulsions.
* Known history of intolerance or hypersensitivity to DEX.
* Any other condition that, in the opinion of the investigator(s), would adversely affect the subject's ability to complete the study or its measure.
* Suicide attempt occurred during time of ECT commencement decision, otherwise, active suicidal intent in MDD with the absence of psychotic symptoms is not an exclusion criterion.
* Able to participate in the trial and adhere to the clinical trial protocol.
* Can provide a written informed consent to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 1-3 WEEKS
  Change in MADRS (Montgomery-Asberg Depression Rating Scale) scores from baseline.
  * Response: >50% reduction in MADRS from baseline and a score <22
  * Remission: MADRS ≤ 10

IPD SHARING:
Plan to Share IPD: Undecided